CLINICAL TRIAL: NCT02011412
Title: The Intermountain Risk Score's Association With Mortality Prediction in Trauma Patients
Brief Title: Intermountain Risk Score and Trauma
Status: Completed | Type: Observational
Sponsor: Intermountain Health Care, Inc. (Other)
Responsible Party: Principal Investigator, Sarah Majercik, Sarah Majercik MD, MBA, FACS, Division of Trauma and Surgical Critical Care, Intermountain Health Care, Inc.
Other Study IDs: 1024710
Record Dates: First submitted 2013-11-06; First posted 2013-12-13 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Trauma; Injury
Keywords: Trauma; Scoring Systems; Intermountain Risk Score
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Intermountain Risk Score known
- Intermountain Risk Score Unknown

SUMMARY:
The investigators hypothesize that a risk score composed of age, sex, and the components of commonly ordered laboratory panels will be predictive of mortality in trauma patients, and will help improve clinicians' ability to make more accurate mortality predictions at the time of admission.

ELIGIBILITY:
Inclusion Criteria:

* Patient presents to Intermountain Medical Center as a Level I or Level II trauma activation.
* Age ≥18

Exclusion Criteria:

* Patients who are not admitted to the hospital

  1. Patients who expire in the Emergency Department
  2. Patients who are discharged to home from the Emergency Department
* Patients who do not have a complete blood count and basic metabolic profile drawn in the Emergency Department as part of routine clinical care.
* Patients who enter the hospital as "trauma consults." These patients have traumatic injuries, and are often admitted to the trauma service, but the severity of their trauma is not thought to warrant trauma team activation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals who suffer from a traumatic injury and present to the Emergency Department as a Trauma Activation
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2013-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
all cause mortality | 30 days
  To determine whether the Intermountain Risk Score accurately predicts 30 day mortality and one year mortality in trauma patients.
all cause mortality | 1 year
  measure the ability of the Intermountain Risk Score to predict all cause mortality at one year after the traumatic event

SECONDARY OUTCOMES:
experienced clinicians mortality prediction | 30 days
  compare the IMRS to experienced clinicians' ability to predict mortality at 30 days
Experienced Clinicians' mortality prediction | 1 year
  compare the IMRS to experienced clinicians' ability to predict mortality at 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Intermountain Medical Center, Murray, Utah, United States